CLINICAL TRIAL: NCT04917159
Title: Effectiveness of Acceptance and Commitment Therapy on the Health-related Quality of Life in Patients With Chronic Heart Failure and Their Family Caregivers: A Randomized Controlled Trial
Brief Title: Acceptance and Commitment Therapy for Patients With Chronic Heart Failure and Their Caregivers on Their Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PU001
Record Dates: First submitted 2021-05-26; First posted 2021-06-08 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2022-05

CONDITIONS: Chronic Heart Failure
Keywords: Chronic heart failure; Acceptance and Commitment Therapy; Patient-caregiver dyads; Health-related quality of life; Randomized controlled trial
MeSH Terms: interventions — Helium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Group (Experimental): The ACT intervention was structured to take place over one month on a weekly basis via Tencent's VooV platform. Each roughly 2-hour session will consist of a group-based ACT (1.5 hours) and a brief health education talk on CHF self-management (0.5 hours). Each training session will serve about 4-8 dyads. In addition, each participant will receive one set of session handouts on CHF education, ACT skills, and a homework assignment.
  Interventions: Behavioral: ACT (Acceptance and Commitment Therapy) plus brief CHF education
- HE group (Active Comparator): The participants of the control group will receive four weekly 2-hour sessions of structured health education on CHF self-management over four consecutive weeks via Tencent's VooV platform, delivered by a registered nurse. Each session will includea a review of the previous session (except the first session), a CHF education talk and a Q&A section to evaluate the participant's understanding of the key concepts. Each session will be offered to 4-8 patient-caregiver dyads. In addition, each participant will receive session handouts on the main topic related to CHF self-management and homework assignments.
  Interventions: Behavioral: HE (Health Education)

INTERVENTIONS:
Behavioral: ACT (Acceptance and Commitment Therapy) plus brief CHF education — The participants will identify their values and clarify their alternative behavior, exploring their thoughts and feelings, and finding ways to meet their own and their family member's needs. The rational bond between the patient and his/her family caregiver will be emphasized. In addtion, the contents of brief CHF education are based on the latest national clinical practice guideline for CHF, including symptoms monitoring, medication adherence, fluid and salt restriction, smoking cessation, alcohol consumption, and physical activity maintenance.
  Arms: ACT Group
Behavioral: HE (Health Education) — The educational contents are based on the latest national clinical practice guideline for CHF. Besides the basic information on CHF education provided in intervention group, the contents of CHF education also include definition of CHF, epidemiology, diagnosis, comorbidity, and CHF treatment. ACT components are not covered.
  Arms: HE group

SUMMARY:
This study is to examine whether group-based Acceptance and Commitment Therapy in the patient-caregiver dyads with Chronic Heart Failure is effective in improving dyadic health-related quality of life, dyadic psychological symptoms, caregiver burden, the rate of patient's readmission, and patient's self-care behavior in comparison with those dyads receiving health education over three-month post intervention.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) is a complex progressive debilitating illness characterized by high morbidity and mortality with unpredictable course and frequent hospital readmissions. Patients with CHF are often old with comorbid impaired psychosocial functioning, and worse health-related quality of life (HRQoL), which generate unavoidable increased dependence on their family caregivers at home. The family caregivers often bear physical and psychological challenges with declined HRQoL, maintaining interdependent relationships with their care recipient when participating in CHF self-management. Dyadic interventions delivered to the patients along with their family caregivers are successful to facilitate patients' self-management to reduce patients' hospital readmission rates and improve HRQoL for both patients and their caregivers post-discharge in the context of chronic disease management. However, little attention has been paid to this vulnerable group. It is noteworthy that a transdiagnostic psychological approach, Acceptance and Commitment Therapy (ACT), aiming to promote psychological flexibility, has demonstrated an ability to break through the psychological barriers to meaningful living among clinical and non-clinical populations. Existing evidence shows promising improvements of ACT on HRQoL in both patients with chronic illness and the family caregivers of the patients with childhood illness. Such evidence implies that ACT in the patient-caregiver dyads may be beneficial for HRQoL and other health outcomes for both patients with CHF and their family caregivers. However, little has been done to address these concerns in mainland China.

A pilot testing was to evaluate the feasibility of recruiting participants at the clinical setting and the acceptability of group-based ACT to patient-caregiver dyads with CHF. Then, a pragmatic, single-center, two-arm, parallel (in 1:1 ratio) randomized controlled trial (RCT) will be performed to examine the effects of acceptance and commitment therapy in patient-caregiver dyads with CHF. Eligible patient-caregiver dyads will be randomly assigned to either the intervention group or the control group. Assessments will be conducted before the intervention, immediately post-intervention, and 3-month post-intervention by blind outcome assessors. The ACT intervention will be delivered by two facilitators and continually supervised by an experienced ACT researcher.

ELIGIBILITY:
Patient-caregiver dyads will be recruited as units if both are eligible as listed below.

1. Patient

   * Inclusion Criteria:

     * 18 years or older
     * a confirmed diagnosis of Chronic Heart Failure (CHF) according to international guidelines
     * with New York Heart Association (NYHA) functional classification I to III
     * has been hospitalized in the past one year
     * able to nominate a primary family caregiver (if two or more family members where the primary caregivers of the patient, the one who had the highest average contact hours with the patient)
     * can understand and communicate in Chinese
     * can access Tencent VooV Meeting via smartphone for attending the intervention
   * Exclusion Criteria:

     * has a documented medical history of psychiatric illness, dementia, and life-threatening, such as end-stage renal failure, severe pulmonary disease and respiratory disease
     * has cognitive impairment evaluated with a score of 0-2 on the Mini-Cog scale
     * living in a nursing home
2. Caregiver

   * Inclusion Criteria:

     * 18 years or older
     * can understand and communicate in Chinese
     * have been providing care to the patient for more than 14 hours per week for at least three consecutive months
     * can access Tencent VooV Meeting via smartphone for attending the intervention
   * Exclusion Criteria:

     * paid caregivers
     * has a documented medical history of psychiatric illness, dementia, and life-threatening, such as end-stage renal failure, severe pulmonary disease and respiratory disease
     * has cognitive impairment evaluated with a score of 0-2 on the Mini-Cog scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patients' CHF specific health-related quality of life at immediately post-intervention | Baseline and post-intervention immediately
  The short-form Kansas City Cardiomyopathy Questionnaire (KCCQ-12) will be used for patients. KCCQ-12 is a 12-item instrument with a score of 0-100, a lower score indicates a poorer quality of life.
Change from baseline in patients' CHF specific health-related quality of life at 3-month post-intervention | Baseline and three-month post-intervention
  The short-form Kansas City Cardiomyopathy Questionnaire (KCCQ-12) will be used for patients. KCCQ-12 is a 12-item instrument with a score of 0-100, a lower score indicates a poorer quality of life.
Change from baseline in patients' generic health-related quality of life at immediately post-intervention | Baseline and post-intervention immediately
  The five-dimensional descriptive system of the EuroQol Group 5-Dimension questionnaire (EQ-5D-5L) will be used to evaluate generic health-related quality of life for patients. The scores range from less than 0 to 1.0, with higher scores representing higher health utility.
Change from baseline in patients' generic health-related quality of life at three-month post-intervention | Baseline and three-month post-intervention
  The five-dimensional descriptive system of the EuroQol Group 5-Dimension questionnaire (EQ-5D-5L) will be used to evaluate generic health-related quality of life for patients. The scores range from less than 0 to 1.0, with higher scores representing higher health utility.
Change from baseline in caregivers' health-related quality of life at immediately post-intervention | Baseline and post-intervention immediately
  The five-dimensional descriptive system of the EuroQol Group 5-Dimension questionnaire (EQ-5D-5L) will be used to evaluate generic health-related quality of life for caregivers. The scores range from less than 0 to 1.0, with higher scores representing higher health utility.
Change from baseline in caregivers' health-related quality of life at three-month post-intervention | Baseline and three-month post-intervention
  The five-dimensional descriptive system of the EuroQol Group 5-Dimension questionnaire (EQ-5D-5L) will be used to evaluate generic health-related quality of life for caregivers. The scores range from less than 0 to 1.0, with higher scores representing higher health utility.

SECONDARY OUTCOMES:
Change from baseline in patients' unscheduled health service visits due to heart-related problems at immediately post-intervention | Baseline and post-intervention immediately
  Patients' report of the total number of unscheduled readmission and emergency visits due to heart-related problems in either a / public hospital(s) and/or a private hospital(s)
Change from baseline in patients' unscheduled health service visits due to heart-related problems at three-month post-intervention | Baseline and three-month post-intervention
  Patients' report of the total number of unscheduled readmission and emergency visits due to heart-related problems in either a / public hospital(s) and/or a private hospital(s)
Change from baseline in patients' CHF self-care behavior at immediately post-intervention | Baseline and post-intervention immediately
  The European Heart Failure Self-care Behavior Scale (EHFScBS) will be used for patients to evaluate their self-care behavior. EHFScBS is a 12-item 5-point Likert scale with a score ranging from 0 to 60, a lower score represents a higher level of self-care behaviors.
Change from baseline in patients' CHF self-care behavior at immediately post-intervention | Baseline and three-month post-intervention
  The European Heart Failure Self-care Behavior Scale (EHFScBS) will be used for patients to evaluate their self-care behavior. EHFScBS is a 12-item 5-point Likert scale with a score ranging from 0 to 60, a lower score represents a higher level of self-care behaviors.
Change from baseline in patients' smoking status at immediately post-intervention | Baseline and post-intervention immediately
  Patients' report of not having/ having smoked and the estimated amount of cigarette consumed (if applicable) for the past one week.
Change from baseline in patients' smoking status at three-month post-intervention | Baseline and three-month post-intervention
  Patients' report of not having/ having smoked and the estimated amount of cigarette consumed (if applicable) for the past one week.
Change from baseline in patients' alcohol status at immediately post-intervention | Baseline and post-intervention immediately
  Patients' report of not having/ having alcohol drinking and the estimated amount of alcohol consumed (if applicable) for the past one week.
Change from baseline in patients' alcohol status at three-month post-intervention | Baseline and three-month post-intervention
  Patients' report of not having/ having alcohol drinking and the estimated amount of alcohol consumed (if applicable) for the past one week.
Change from baseline in caregivers' perceived care burden at immediately post-intervention | Baseline and post-intervention immediately
  The Zarit Caregiver Burden Interview (ZBI) will be used for caregivers to evaluate perceived care burden. ZBI is a 22-item 5-point Likert scale with a score ranging from 0 to 88, a lower score indicates less care burden.
Change from baseline in caregivers' perceived care burden at three-month post-intervention | Baseline and three-month post-intervention
  The Zarit Caregiver Burden Interview (ZBI) will be used for caregivers to evaluate perceived care burden. ZBI is a 22-item 5-point Likert scale with a score ranging from 0 to 88, a lower score indicates less care burden.
Change from baseline in participants' anxiety symptoms at immediately post-intervention | Baseline and post-intervention immediately
  The General Anxiety Disorder Scale (GAD) will be used for caregivers and patients. The GAD consists of 7 item 4-point Likert scale. The score of each scale ranges from 0 to 21, with a lower score indicating a lower level of anxiety.
Change from baseline in participants' depressive symptoms at immediately post-intervention | Baseline and post-intervention immediately
  The Patient Health Questionaire (PHQ) will be used for caregivers and patients. The PHQ consists of 9 item 4-point Likert scale. The score of each scale ranges from 0 to 27, with a lower score indicating a lower level of depression.
Change from baseline in participants' anxiety symptoms at three-month post-intervention | Baseline and three-month post-intervention
  The General Anxiety Disorder Scale (GAD) will be used for caregivers and patients. The GAD consists of 7 item 4-point Likert scale. The score of each scale ranges from 0 to 21, with a lower score indicating a lower level of anxiety.
Change from baseline in participants' depressive symptoms at three-month post-intervention | Baseline and three-month post-intervention
  The Patient Health Questionaire (PHQ) will be used for caregivers and patients. The PHQ consists of 9 item 4-point Likert scale. The score of each scale ranges from 0 to 27, with a lower score indicating a lower level of depression.
Change from baseline in participants' perspective taking at immediately post-intervention | Baseline and post-intervention immediately
  The perspective taking subscale from the Interpersonall Reactivity Index (IRI) will be used for caregivers and patients. Chinese version of the perspective taking subscale is a 5-item 5-point Likert scale with a score ranging from 5 to 25, a lower score represents a lower tendency for perspective taking.
Change from baseline in participants' perspective taking at three-month post-intervention | Baseline and three-month post-intervention
  The perspective taking subscale from the Interpersonall Reactivity Index (IRI) will be used for caregivers and patients. Chinese version of the perspective taking subscale is a 5-item 5-point Likert scale with a score ranging from 5 to 25, a lower score represents a lower tendency for perspective taking.
Change from baseline in participants' psychological flexibility at immediately post-intervention | Baseline and post-intervention immediately
  The Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT) will be used for caregivers and patients.CompACT is an 18-item 5-point Likert scale with a score ranging from 18 to 90, a lower score represents a lower level of psychological flexibility.
Change from baseline in participants' psychological flexibility at three-month post-intervention | Baseline and three-month post-intervention
  The Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT) will be used for caregivers and patients.CompACT is an 18-item 5-point Likert scale with a score ranging from 18 to 90, a lower score represents a lower level of psychological flexibility.
Change from baseline in participants' relationship functioning at immediately post-intervention | Baseline and post-intervention immediately
  The Dyadic Adjustment Scale-7(DAS-7) will be used for caregivers and patients.DAS-7 is a 7-item 6-point Likert scale with a score ranging from 0 to 36, a lower score represents less positive relationship quality.
Change from baseline in participants' relationship functioning at three-month post-intervention | Baseline and three-month post-intervention
  The Dyadic Adjustment Scale-7(DAS-7) will be used for caregivers and patients.DAS-7 is a 7-item 6-point Likert scale with a score ranging from 0 to 36, a lower score represents less positive relationship quality.
Change from baseline in participants' generic health-related quality of life at immediately post-intervention | Baseline and post-intervention immediately
  The visual analog scale (VAS) of EuroQol Group 5-Dimension questionnaire (EQ-5D-5L) will be used to evaluate participants' perceived health, the score ranges from 0 to 100 with 100 being better.
Change from baseline in participants' generic health-related quality of life at three-month post-intervention | Baseline and three-month post-intervention
  The visual analog scale (VAS) of EuroQol Group 5-Dimension questionnaire (EQ-5D-5L) will be used to evaluate participants' perceived health, the score ranges from 0 to 100 with 100 being better.
Change from baseline in participants' self-compassion at immediately post-intervention | Baseline and post-intervention immediately
  The Self-compassion Scale (SCS) will be used for caregivers and patients.SCS is an 12-item 5-point Likert scale with a score ranging from 12 to 60, a lower score represents a lower level of self-compassion.
Change from baseline in participants' self-compassion at three-month post-intervention | Baseline and three-month post-intervention
  The Self-compassion Scale (SCS) will be used for caregivers and patients.SCS is an 12-item 5-point Likert scale with a score ranging from 12 to 60, a lower score represents a lower level of self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Yim Wah Mak, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- Taihe Hospital, Shiyan, Hubei, China

REFERENCES:
- [Derived] Zhang X, Ho GWK, Mak YW. Effectiveness of a videoconferencing group-based dyad acceptance and commitment therapy on the quality of life of chronic heart failure patients and their family caregivers: A study protocol for a randomized controlled trial. PLoS One. 2024 Apr 18;19(4):e0298178. doi: 10.1371/journal.pone.0298178. eCollection 2024. PMID 38635558